CLINICAL TRIAL: NCT02958865
Title: A PHASE 2B, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, PARALLEL GROUP, DOSE RANGING STUDY OF ORAL PF-06651600 AND PF-06700841 AS INDUCTION AND CHRONIC THERAPY IN SUBJECTS WITH MODERATE TO SEVERE ULCERATIVE COLITIS
Brief Title: Study to Compare Oral PF-06651600, PF-06700841 and Placebo in Subjects With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B7981005; VIBRATO (Other: Alias Study Number); 2016-003708-29 (EudraCT Number)
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Ulcerative Colitis
Keywords: Mayo score
MeSH Terms: conditions — Colitis, Ulcerative | interventions — PF-06651600; PF-06700841

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- PF-06651600 Drug Dose Level 1 (Experimental): Delivered orally for 8 weeks
  Interventions: Drug: PF-06651600 or Placebo
- PF-06651600 Drug Dose Level 2 (Experimental): Delivered orally for 8 weeks
  Interventions: Drug: PF-06651600 or Placebo
- PF-06651600 Drug Dose Level 3 (Experimental): Delivered orally for 8 weeks.
  Interventions: Drug: PF-06651600 or Placebo
- PF-06651600 Placebo (Placebo Comparator): Delivered orally for 8 weeks.
  Interventions: Drug: PF-06651600 or Placebo
- PF-06700841 Drug Dose Level 1 (Experimental): Delivered orally for 8 weeks
  Interventions: Drug: PF-06700841 or Placebo
- PF-06700841 Drug Dose Level 2 (Experimental): Delivered orally for 8 weeks.
  Interventions: Drug: PF-06700841 or Placebo
- PF-06700841 Drug Dose Level 3 (Experimental): Delivered orally for 8 weeks.
  Interventions: Drug: PF-06700841 or Placebo
- PF-06700841 Placebo (Placebo Comparator): Delivered orally for 8 weeks.
  Interventions: Drug: PF-06700841 or Placebo
- PF-06651600 Drug Dose Level 4 (Experimental): Delivered orally for 24 weeks.
  Interventions: Drug: PF-06651600
- PF-06700841 Drug Dose Level 4 (Experimental): Delivered orally for 24 weeks.
  Interventions: Drug: PF-06700841

INTERVENTIONS:
Drug: PF-06651600 or Placebo — Delivered orally for 8 weeks.
  Arms: PF-06651600 Drug Dose Level 1; PF-06651600 Drug Dose Level 2; PF-06651600 Drug Dose Level 3; PF-06651600 Placebo
Drug: PF-06700841 or Placebo — Delivered orally for 8 weeks.
  Arms: PF-06700841 Drug Dose Level 1; PF-06700841 Drug Dose Level 2; PF-06700841 Drug Dose Level 3; PF-06700841 Placebo
Drug: PF-06700841 — Delivered orally for 24 weeks.
  Arms: PF-06700841 Drug Dose Level 4
Drug: PF-06651600 — Delivered orally for 24 weeks.
  Arms: PF-06651600 Drug Dose Level 4

SUMMARY:
The purpose of this study is to determine whether PF-06651600 and PF-06700841 are effective in treatment of moderate to severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis for greater than/equal to 3 months.
* Moderate to severe active ulcerative colitis
* Inadequate response to, loss of response to, or intolerance to at least one conventional therapy for UC.

Exclusion Criteria:

* Pregnant or breastfeeding
* Clinical findings suggestive of Crohn's Disease
* History of bowel surgery within 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (186):
- United States (58):
  - Dothan Surgery Center, Dothan, Alabama
  - Gut P.C., dba Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Long Beach Clinical Trials Services Inc., Long Beach, California
  - Southern California Research Institute Medical Group/West Gastroenterology Medical Group/Airport En-, Los Angeles, California
  - Clinical Application Laboratories, INC., San Diego, California
  - San Diego Endoscopy Center, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Front Range Endoscopy Center, Colorado Springs, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Bristol Hospital, Bristol, Connecticut
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Central Connecticut Endoscopy Center, Plainville, Connecticut
  - West Coast Endoscopy Center, Clearwater, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Millenia Surgery Center, Orlando, Florida
  - HMD Research LLC, Orlando, Florida
  - Orlando Gastroenterology, PA, Orlando, Florida
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland
  - Feldman ENT, Chevy Chase, Maryland
  - MGG Group Co. Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Cascades Endoscopy Center, Columbia, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Concorde medical Group, PLLC, New York, New York
  - Kips Bay Endoscopy Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - NYU Clinical Cancer Center, New York, New York
  - NYU Langone Medical Center, New York, New York
  - NYU Medical Science Building, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College, New York, New York
  - New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - UNC Hospitals Endoscopy Center at Meadowmont, Chapel Hill, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Gastro One, Germantown, Tennessee
  - Parkland Health and Hospital System, Dallas, Texas
  - UT Southwestern Medical Center - CRU Aston, Dallas, Texas
  - UT Southwestern Medical Center-Clements University Hospital, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine- Baylor Medical Center, Houston, Texas
  - Baylor St. Luke's Medical Center Endoscopy-McNair Campus, Houston, Texas
  - Gulf Coast Research Group, Houston, Texas
  - Lonestar Endoscopy, LLP, Keller, Texas
  - Sagact, Pllc., San Antonio, Texas
  - Sagact, Pllc, San Antonio, Texas
  - Lonestar Endoscopy, LLP, Southlake, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Verity Research, Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - University of Washington, Seattle, Washington
- AKH Wien Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Bulgaria (9):
  - "Medical Center-1- Sevlievo" EOOD, Sevlievo, Gabrovo
  - "MHAT-Blagoevgrad" AD, Blagoevgrad
  - MHAT Dobrich AD, Dobrich
  - MC Hipocrat-2000 OOD, Haskovo
  - MHAT Prof. Dr. Paraskev Stoyanov AD, Lovech
  - Medical Center Vitadar Consult OOD, Rousse
  - SHATPPD dr. Dimitar Gramatikov - Ruse EOOD, Rousse
  - "MC Asklepion - researches in human medicine"" EOOD, Sofia
  - "Acibadem City Clinic UMHAT" EOOD, Sofia
- Czechia (4):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Slany, p.o., Slaný
  - Nemocnice Strakonice, a.s., interni oddeleni, Strakonice
- Denmark (4):
  - Nordsjaellands Hospital Frederikssund, Frederikssund
  - Nordsjaellands Hospital Hilleroed, Hilleroed
  - Amager og Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense
- Georgia (2):
  - Research institute of Clinical Medicine, Tbilisi
  - The First University Clinic of TSMU, Tbilisi
- Germany (8):
  - Paian MED Research GmbH, Berlin
  - Gastrostudien GbR, Berlin
  - Krankenhaus Waldfriede e.V., Berlin
  - MVZ Dachau - Patientenzentrum, Dachau
  - MVZ Dachau, Dachau
  - Asklepios Westklinikum Hamburg, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Eugastro GmbH, Leipzig
- Hungary (6):
  - Bekes Megyei Kozponti Korhaz, Rethy Pal Tagkorhaz, Békéscsaba
  - Semmelweis Egyetem, II. Belgyogyaszati Klinika, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak I. Belgyogyaszati Gasztroenterologiai Osztaly, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Javorszky Odon Korhaz, Gasztroenterologia, Vác
- Israel (4):
  - Clalit Health Services, Bat Yam
  - Shaare Zedek Medical Center, Jerusalem
  - Diabetes and Endocrinology Unit, Tel Aviv
  - Migdal Hamea Clinic, Tel Aviv
- Italy (10):
  - IRCCS Saverio De Bellis, Castellana Grotte, BARI
  - AOU Sant'Orsola-Malpighi, Bologna, BO
  - A.O.U. Policlinico G. Martino, Messina, ME
  - Istituto Clinico Humanitas, Rozzano, Milan (MI)
  - ASST Rhodense - Ospedale di Circolo di Rho, Rho, Milano (MI)
  - Azienda Ospedaliero Universitaria Pisana, Pisa, PI
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - AOU Policlinico di Modena, Modena
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Sanitaria Universitaria Integrata Udine, Udine
- Poland (14):
  - SPZOZ Wojewodzki Szpital Zespolony im. Jedrzeja Sniadeckiego w Bialymstoku, Bialystok
  - ETG Kielce, Kielce
  - Gastromed Sp. z o.o., Lublin
  - Ai Centrum Medyczne Sp. Z O.O. Sp.K., Poznan
  - KO-MED Centra Kliniczne Pulawy, Puławy
  - ENDOSKOPIA Sp. z o. o., Sopot
  - H-T. Centrum Medyczne, Tychy
  - Centrum Zdrowia MDM, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Melita Medical Sp z o.o., Wroclaw
  - Centrum Badan Klinicznych, Osrodek Badan Wczesnej Fazy, Wroclaw
  - Lexmedica, Wroclaw
  - EMC Instytut Medyczny S.A., Szpital Specjalistyczny EuroMediCare z Przychodnia, Wroclaw
  - Centrum Diagnostyczno-Lecznicze Barska Sp. z o. o., Włocławek
- Romania (3):
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila" Bucuresti, Bucharest, Sector 1,
  - S.C. Cabinet Particular Policlinic Algomed SRL, Timișoara, Timiș County
  - Spitalul Clinic Colentina, Sectia de Gastroenterologie, Bucharest
- Russia (15):
  - LLC "Olla-Med", Moscow
  - FSAEI HE I.M.Sechenov 1st Moscow State Medical University of the MoH of the RF (Sechenov University), Moscow
  - Limited Liability Company "Medicinsky Center SibNovoMed", Novosibirsk
  - LLC Novosibirskiy Gastrocentr, Novosibirsk
  - Novosibirskiy Gastrocenter, Novosibirsk
  - Federal State Budgetary Scientific Institution, Novosibirsk
  - FGBOU VO OmGMU Minzdrava Rossii, Omsk
  - FSBEI HE "Rostov State Medical University" of the Ministry of Healthcare of the Russian Federation, Rostov-on-Don
  - State Budgetary Institution of Ryazan Region "Regional Clinical Hospital", Ryazan
  - RIAT Limited Liability Company (RIAT LLC), Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution, Saint Petersburg
  - Medical University REAVIZ, Samara
  - Private Healthcare Institution "Clinical Hospital "RZhD-Medicina" City Samara", Samara
  - LLC Medical Company Hepatolog, Samara
  - State Budgetary Institution of Healthcare Yaroslavl Regional Clinical Hospital, Yaroslavl
- Serbia (7):
  - Clinical Hospital Centre Zvezdara Clinic for Internal Diseases, Belgrade
  - Clinical Hospital Centre Bezanijska Kosa Clinic for Internal Medicine, Belgrade
  - Clinical Centre of Kragujevac, Kragujevac
  - Clinical Centre of Nis, Clinic for Gastroenterology and Hepatology, Niš
  - General Hospital Subotica, Subotica
  - Clinical Hospital Center Zemun, Zemun, Belgrade
  - General Hospital "Djordje Joanovic", Zrenjanin
- Slovakia (4):
  - Abawi spol. s r.o, Bratislava
  - KM Management spol. s.r.o., Nitra
  - MUDr. Frantisek Horvath Gastroenterologia, Šahy
  - ENDOMED, s.r.o., Vranov nad Topľou
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (7):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (12):
  - Ankara Universitesi Tip Fakultesi, Ibn-i Sina Hastanesi, Ic Hastaliklari Anabilim Dali,, Ankara
  - Ankara Universitesi Tip Fakultesi, Ibn-i-Sina Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tıp Fakultesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Bulent Ecevit Universitesi Tip Fakultesi, Kozlu Zonguldak
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin
  - Bulent Ecevit Universitesi Tip Fakultesi, Zonguldak
- Ukraine (14):
  - Regional Consultative Polyclinic, Chernivtsi
  - Regional Municipal Institution "Chernivtsi Regional Clinical Hospital", gastroenterology department,, Chernivtsi
  - MNCECCH No.2 n.a. PROF O.O. SHALIMOV of KHARKIV CITY COUNCIL, Kharkiv
  - Municipal Institution "Kherson City Clinical Hospital n.a. Afanasiy and Olga Tropiny", Kherson
  - Private Enterprise of Private Manufacturing Company "Acinus", Medical and Diagnostic Center, Kropyvnytskyi
  - Kyiv Municipal Clinical Hospital #18, Proctology Department, Kyiv
  - Medical Center "Universal clinic Oberig" of "Kapital" LLC, Gastro center, Kyiv
  - Lviv clinical hospital on Railway Transport of Health Care Center branch of PJSC Ukrainian Railway, Lviv
  - Municipal Non-Profit Enterprise "Lviv Clinical Emergency Care Hospital", Lviv
  - Municipal Institution "Odesa Regional Clinical Hospital", Odesa
  - Municipal Institution of Ternopil regional council Ternopil University Hospital, Ternopil
  - Municipal Institution "Uzhgorod Regional Hospital", Uzhhorod
  - Zakarpattia Regional Clinical Hospital n.a. A. Novak,, Uzhhorod
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrohov, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hassan-Zahraee M, Ye Z, Xi L, Dushin E, Lee J, Romatowski J, Leszczyszyn J, Danese S, Sandborn WJ, Banfield C, Gale JD, Peeva E, Longman RS, Hyde CL, Hung KE. Baseline Serum and Stool Microbiome Biomarkers Predict Clinical Efficacy and Tissue Molecular Response After Ritlecitinib Induction Therapy in Ulcerative Colitis. J Crohns Colitis. 2024 Sep 3;18(9):1361-1370. doi: 10.1093/ecco-jcc/jjad213. PMID 38141256
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Sandborn WJ, Danese S, Leszczyszyn J, Romatowski J, Altintas E, Peeva E, Hassan-Zahraee M, Vincent MS, Reddy PS, Banfield C, Salganik M, Banerjee A, Gale JD, Hung KE. Oral Ritlecitinib and Brepocitinib for Moderate-to-Severe Ulcerative Colitis: Results From a Randomized, Phase 2b Study. Clin Gastroenterol Hepatol. 2023 Sep;21(10):2616-2628.e7. doi: 10.1016/j.cgh.2022.12.029. Epub 2023 Jan 6. PMID 36623678
- [Derived] Fensome A, Ambler CM, Arnold E, Banker ME, Brown MF, Chrencik J, Clark JD, Dowty ME, Efremov IV, Flick A, Gerstenberger BS, Gopalsamy A, Hayward MM, Hegen M, Hollingshead BD, Jussif J, Knafels JD, Limburg DC, Lin D, Lin TH, Pierce BS, Saiah E, Sharma R, Symanowicz PT, Telliez JB, Trujillo JI, Vajdos FF, Vincent F, Wan ZK, Xing L, Yang X, Yang X, Zhang L. Dual Inhibition of TYK2 and JAK1 for the Treatment of Autoimmune Diseases: Discovery of (( S)-2,2-Difluorocyclopropyl)((1 R,5 S)-3-(2-((1-methyl-1 H-pyrazol-4-yl)amino)pyrimidin-4-yl)-3,8-diazabicyclo[3.2.1]octan-8-yl)methanone (PF-06700841). J Med Chem. 2018 Oct 11;61(19):8597-8612. doi: 10.1021/acs.jmedchem.8b00917. Epub 2018 Aug 16. PMID 30113844
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a screening period of up to 6 weeks, an 8-week double-blind induction period, and an additional 24-week open-label active chronic dosing period followed by a 4-week follow up period after the last dose of investigational product.
Pre-assignment Details: A total of 319 participants were randomized and 317 participants were treated.
Groups:
- Placebo (Induction): The placebo was administered orally once daily (QD) from Day 1 to Week 8.
- PF-06651600 20 mg (Induction): PF-06651600 tablet was administered orally at 20 mg QD from Day 1 to Week 8.
- PF-06651600 70 mg (Induction): PF-06651600 tablet was administered orally at 70 mg QD from Day 1 to Week 8.
- PF-06651600 200 mg (Induction): PF-06651600 tablet was administered orally at 200 mg QD from Day 1 to Week 8.
- PF-06700841 10 mg (Induction): PF-06700841 tablet was administered orally at 10 mg QD from Day 1 to Week 8.
- PF-06700841 30 mg (Induction): PF-06700841 tablet was administered orally at 30 mg QD from Day 1 to Week 8.
- PF-06700841 60 mg (Induction): PF-06700841 tablet was administered orally at 60 mg QD from Day 1 to Week 8.
- PF-06651600 200 mg -> PF-06651600 50 mg: PF-06651600 tablet was administered orally at 200 mg QD from Day 1 to Week 8 and at 50 mg QD from Week 9 to Week 32.
- PF-06651600 70 mg -> PF-06651600 50 mg: PF-06651600 tablet was administered orally at 70 mg QD from Day 1 to Week 8 and at 50 mg QD from Week 9 to Week 32.
- PF-06651600 20 mg -> PF-06651600 50 mg: PF-06651600 tablet was administered orally at 20 mg QD from Day 1 to Week 8 and at 50 mg QD from Week 9 to Week 32.
- Placebo -> PF-06651600 50 mg: The placebo was administered orally QD from Day 1 to Week 8 and PF-06651600 was administered at 50 mg QD from Week 9 to Week 32.
- PF-06700841 60 mg -> PF-06700841 30 mg: PF-06700841 tablet was administered orally at 60 mg QD from Day 1 to Week 8 and at 30 mg QD from Week 9 to Week 32.
- PF-06700841 30 mg -> PF-06700841 30 mg: PF-06700841 tablet was administered orally at 30 mg QD from Day 1 to Week 8 and at 30 mg QD from Week 9 to Week 32.
- PF-06700841 10 mg -> PF-06700841 30 mg: PF-06700841 tablet was administered orally at 10 mg QD from Day 1 to Week 8 and at 30 mg QD from Week 9 to Week 32.
- Placebo -> PF-06700841 30 mg: The placebo was administered orally from Day 1 to Week 8 and PF-06700841 was administered orally at 30 mg QD from Week 9 to Week 32.
- Pooling Placebo During Chronic: The placebo was administered orally QD from Week 9 to Week 32 regardless of what was administered from Day 1 to Week 8.
Period: Induction Period (Day 1 to Week 8)
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction) | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Started | 25 | 51 | 49 | 50 | 48 | 47 | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 21 | 44 | 43 | 41 | 45 | 43 | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 7 | 6 | 9 | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 0 | 5 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer meeting eligibility criteria | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Chronic Period (Week 8 to Week 32)
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction) | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 36 | 39 | 10 | 38 | 37 | 39 | 9 | 37
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 33 | 33 | 10 | 31 | 26 | 31 | 5 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 6 | 0 | 7 | 11 | 8 | 4 | 17
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 4 | 1 | 1 | 5
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 5 | 0 | 2 | 0 | 8
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 3 | 3 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — No longer meeting eligibility criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of PF-06651600, PF-06700841, or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction) | Total
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47 | 317
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (15.45) | 41.3 (14.03) | 40.2 (13.31) | 37.3 (15.67) | 40.8 (13.04) | 40.9 (13.03) | 40.3 (12.80) | 40.3 (13.79)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 13 | 31 | 30 | 36 | 31 | 25 | 30 | 196
  45-64 years | 10 | 16 | 18 | 10 | 16 | 22 | 16 | 108
  >=65 years | 2 | 4 | 1 | 4 | 1 | 0 | 1 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 25 | 18 | 18 | 24 | 22 | 135
  Male | 14 | 34 | 24 | 32 | 30 | 23 | 25 | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 46 | 46 | 48 | 44 | 44 | 45 | 295
  Black or African American | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 6
  Asian | 1 | 3 | 1 | 0 | 3 | 3 | 0 | 11
  Other (not specified) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Mayo Score at Week 8 (Induction Period)
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicates more severe disease activity and lower score denotes improvement of disease activity as measured by the total Mayo score.
Time Frame: Week 8
Population: The intent-to-treat (ITT) analysis set which included all randomized participants who received at least 1 dose of investigational product or placebo.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Units on a scale | 7.88 [6.95 to 8.81] | 5.85 [5.18 to 6.51] | 4.00 [3.33 to 4.67] | 3.27 [2.58 to 3.96] | 6.08 [5.43 to 6.74] | 5.60 [4.93 to 6.27] | 4.67 [4.01 to 5.33]
Statistical Analysis 1: Comparison: Placebo (Induction) vs PF-06651600 20 mg (Induction); The null hypothesis was that the there was no difference between the distributions of the total Mayo score at Week 8 between the pooled placebo group and active arm. The treatment arm was declared efficacious if an upper limit of 2-sided 90% confidence interval for the treatment effect was below zero; Test type: Superiority; p = 0.0017, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = -2.03, 90% CI 2-sided [-3.17 to -0.89], Standard Error of Mean 0.69
Statistical Analysis 2: Comparison: Placebo (Induction) vs PF-06651600 70 mg (Induction); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = -3.88, 90% CI 2-sided [-5.01 to -2.74], Standard Error of Mean 0.69
Statistical Analysis 3: Comparison: Placebo (Induction) vs PF-06651600 200 mg (Induction); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = -4.61, 90% CI 2-sided [-5.76 to -3.46], Standard Error of Mean 0.70
Statistical Analysis 4: Comparison: Placebo (Induction) vs PF-06700841 10 mg (Induction); The null hypothesis was that the there is no difference between the distributions of the total Mayo score at Week 8 between the pooled placebo group and active arm. The treatment arm is declared efficacious if an upper limit of 2-sided 90% confidence interval for the treatment effect is below zero; Test type: Superiority; p = 0.0045, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = -1.79, 90% CI 2-sided [-2.92 to -0.67], Standard Error of Mean 0.68
Statistical Analysis 5: Comparison: Placebo (Induction) vs PF-06700841 30 mg (Induction); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0005, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = -2.28, 90% CI 2-sided [-3.41 to -1.14], Standard Error of Mean 0.69
Statistical Analysis 6: Comparison: Placebo (Induction) vs PF-06700841 60 mg (Induction); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = -3.21, 90% CI 2-sided [-4.34 to -2.08], Standard Error of Mean 0.69

2. Secondary Outcome: Number of Participants With AEs, SAEs and Discontinuation Due to AEs (Chronic Period)
Description: An AE was an untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes: death, life-threatening experience, initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. All AEs mentioned below are treatment-emergent AEs.
Time Frame: From Week 8 up to Week 32
Population: The safety analysis set was defined as those participants who received at least one dose of PF-06651600, PF-06700841, or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo -> PF-06651600 50 mg: mg The placebo was administered orally from Day 1 to Week 8 and PF-06651600 at 50 mg QD from Week 9 to Week 32.
- Pooling Placebo During Chronic: The placebo was administered orally from Week 9 to Week 32 regardless of what was administered from Day 1 to Week 8.
Arm/Group | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Number analyzed (Participants) | 35 | 36 | 39 | 10 | 38 | 37 | 39 | 9 | 37
Participants
  Participants with AEs | 18 | 27 | 18 | 8 | 21 | 23 | 26 | 4 | 18
  Participants with SAEs | 3 | 1 | 1 | 0 | 2 | 4 | 2 | 0 | 0
  Participants discontinued from study due to AEs | 1 | 1 | 3 | 1 | 1 | 4 | 1 | 1 | 6

3. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Chronic Period)
Description: The number of participants with a laboratory abnormality meeting the pre-specified criteria defined in the study protocol while on study treatment or during lag time are reported here. Baseline is defined as the last measurement prior to receiving study treatment. Laboratory data included hematology test, serum chemistry test, C-creative protein and viral surveillance.
Time Frame: From Week 8 to Week 32
Population: The participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo -> PF-06651600 50 mg: The placebo was administered orally from Day 1 to Week 8 and PF-06651600 at 50 mg QD from Week 9 to Week 32.
Arm/Group | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 37
Participants | 27 | 31 | 33 | 8 | 29 | 27 | 28 | 8 | 23

4. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities-hematology (Chronic Period)
Description: The number of participants with a laboratory abnormality meeting specified criteria while on study treatment or during lag time are reported here. Baseline is defined as the last measurement prior to receiving study treatment. The list of hematology test parameters were as follows: hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils (absolute, Abs), eosinophils (Abs), monocytes (Abs), basophils (Abs), lymphocytes (Abs), prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT), and reticulocytes (% and Abs). Percentages are displayed for the laboratory tests having a category with greater or equal to 1 evaluable participant.
Time Frame: From Week 8 to Week 32
Population: Number of Participants Analyzed: the participants who received at least one dose of PF-06651600, PF-06700841, or placebo. Number Analyzed: the participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Number analyzed (Participants) | 35 | 36 | 39 | 10 | 38 | 37 | 39 | 9 | 37
Participants
  Hemoglobin (g/dL) <0.8× LLN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Hemoglobin (g/dL) <0.8× LLN | 2 | 2 | 1 | 1 | 3 | 3 | 6 | 2 | 3
  Hematocrit (%) <0.8× LLN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Hematocrit (%) <0.8× LLN | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 2
  Erythrocytes (10^6/mm^3) <0.8× LLN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Erythrocytes (10^6/mm^3) <0.8× LLN | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1
  Reticulocytes (Abs) (10^3/mm^3) >1.5× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 36 | 39 | 9 | 36
  Reticulocytes (Abs) (10^3/mm^3) >1.5× ULN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes Mean Corpuscular Volume (10^-15L) <0.9× LLN: number analyzed (Participants) | 3 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 0
  Erythrocytes Mean Corpuscular Volume (10^-15L) <0.9× LLN | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Platelets (10^3/mm^3) >1.75× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Platelets (10^3/mm^3) >1.75× ULN | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 2
  Reticulocytes/Erythrocytes (%) >1.5× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 36 | 39 | 9 | 36
  Reticulocytes/Erythrocytes (%) >1.5× ULN | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 1
  Leukocytes (10^3/mm^3) >1.5× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Leukocytes (10^3/mm^3) >1.5× ULN | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Lymphocytes (Abs) (10^3/mm^3) <0.8× LLN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Lymphocytes (Abs) (10^3/mm^3) <0.8× LLN | 7 | 6 | 6 | 1 | 0 | 0 | 3 | 0 | 3
  Lymphocytes (Abs) (10^3/mm^3) >1.2× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Lymphocytes (Abs) (10^3/mm^3) >1.2× ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophils (Abs) (10^3/mm^3) <0.8× LLN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Neutrophils (Abs) (10^3/mm^3) <0.8× LLN | 1 | 2 | 0 | 0 | 3 | 1 | 2 | 1 | 1
  Neutrophils (Abs) (10^3/mm^3) >1.2× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Neutrophils (Abs) (10^3/mm^3) >1.2× ULN | 3 | 8 | 11 | 1 | 8 | 6 | 6 | 3 | 6
  Basophils (Abs) (10^3/mm^3) >1.2× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Basophils (Abs) (10^3/mm^3) >1.2× ULN | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
  Eosinophils (Abs) (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Eosinophils (Abs) (10^3/mm^3) >1.2x ULN | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2
  Monocytes (Abs) (10^3/mm^3) >1.2× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Monocytes (Abs) (10^3/mm^3) >1.2× ULN | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
  Activated PTT (second) >1.1× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Activated PTT (second) >1.1× ULN | 0 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  PT (second) >1.1× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  PT (second) >1.1× ULN | 2 | 3 | 2 | 0 | 2 | 2 | 0 | 0 | 0
  Prothrombin INR >1.1× ULN: number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 36
  Prothrombin INR >1.1× ULN | 2 | 3 | 2 | 0 | 2 | 1 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Vital Signs Data (Chronic Period)
Description: The vital signs data included the single sitting blood pressure, pulse rate and temperature. The criteria of vital sign abnormality are indicated below.
Time Frame: From Week 8 to Week 32
Population: The participants evaluated against the criteria during the chronic period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Number analyzed (Participants) | 35 | 35 | 39 | 10 | 38 | 37 | 39 | 9 | 37
Participants
  Sitting Systolic Blood Pressure Value <90 mmHg | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Sitting Systolic Blood Pressure Change ≥30 mmHg Increase | 0 | 3 | 4 | 0 | 3 | 2 | 3 | 0 | 3
  Sitting Systolic Blood Pressure Change ≥30 mmHg Decrease | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Sitting Diastolic Blood Pressure Value <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting Diastolic Blood Pressure Change ≥20 mmHg Increase | 0 | 1 | 6 | 1 | 4 | 2 | 1 | 1 | 1
  Sitting Diastolic Blood Pressure Change ≥20 mmHg Decrease | 2 | 4 | 5 | 0 | 2 | 3 | 1 | 0 | 2
  Sitting Pulse Rate Value <40 beat per minute (bpm) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting Pulse Rate Value >120 bpm | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal ECG Findings (Chronic Period)
Description: The number of participants with abnormal ECG findings during the chronic period (from Week 9 to Week 32) are reported below.
Time Frame: Week 8 to Week 32
Population: The participants evaluated against the criteria during the chronic period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Number analyzed (Participants) | 35 | 36 | 39 | 10 | 38 | 37 | 36 | 9 | 37
Participants
  Abnormal, not clinically significant | 3 | 6 | 2 | 1 | 1 | 2 | 4 | 2 | 4
  Abnormal, clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Serious Infections (Chronic Period)
Description: Serious infections was defined as any infection (for example, viral, bacterial, and fungal) requiring hospitalization or parenteral antimicrobials.
Time Frame: Week 8 to Week 32
Population: The participants who received at least one dose of PF-06651600, PF-06700841, or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Number analyzed (Participants) | 35 | 36 | 39 | 10 | 38 | 37 | 39 | 9 | 37
Participants
  COVID-19 pneumonia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Viral infection | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities-clinical Chemistry (Chronic Period)
Description: The number of participants with a laboratory abnormality meeting specified criteria while on study treatment or during lag time are reported here. Baseline is defined as the last measurement prior to receiving study treatment. The list of serum chemistry test parameters were as follows: blood urea nitrogen, creatinine, cystatin C, glucose, calcium, sodium, potassium, gamma glutamyl transferase, chloride, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, direct bilirubin, alkaline phosphatase, uric acid, albumin, total protein, creatine kinase (CK), total cholesterol, triglycerides, high-density lipoproteins (HDL), and low-density lipoprotein (LDL).
Time Frame: Week 8 to Week 32
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Number analyzed (Participants) | 35 | 36 | 39 | 10 | 38 | 37 | 39 | 9 | 37
Participants
  Bilirubin (mg/dL) >1.5 x ULN | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
  Direct Bilirubin (mg/dL) >1.5 x ULN: number analyzed (Participants) | 3 | 3 | 6 | 1 | 6 | 4 | 4 | 0 | 4
  Direct Bilirubin (mg/dL) >1.5 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin (mg/dL) >1.5 x ULN: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2 | 0 | 2 | 0 | 1
  Indirect Bilirubin (mg/dL) >1.5 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L) >3.0 x ULN | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) >3.0 x ULN | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
  Gamma Glutamyl Transferase (U/L) >3.0 x ULN: number analyzed (Participants) | 2 | 2 | 2 | 0 | 2 | 1 | 2 | 0 | 1
  Gamma Glutamyl Transferase (U/L) >3.0 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L) >3.0 x ULN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Protein (g/dL) <0.8 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein (g/dL) >1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) <0.8 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) >1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen (mg/dL) >1.3 x ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) >1.3 x ULN | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Urate (mg/dL) >1.2 x ULN | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  HDL Cholesterol (mg/dL) <0.8 x LLN | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LDL Cholesterol (mg/dL) >1.2 x ULN | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0
  Triglycerides (mg/dL) >1.3 x ULN | 3 | 2 | 1 | 0 | 2 | 2 | 1 | 0 | 1
  Sodium (Meq/L) <0.95 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium (Meq/L) >1.05 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (Meq/L) <0.9 x LLN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Potassium (Meq/L) >1.1 x ULN | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Chloride (Meq/L) <0.9 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride (Meq/L) >1.1 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) <0.9 x LLN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Calcium (mg/dL) >1.1 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) <0.6 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) >1.5 x ULN | 1 | 3 | 3 | 0 | 1 | 2 | 0 | 0 | 0
  Hemoglobin A1C (%) >1.3 x ULN: number analyzed (Participants) | 3 | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 2
  Hemoglobin A1C (%) >1.3 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatine Kinase (U/L) >2.0 x ULN | 1 | 3 | 2 | 1 | 3 | 10 | 2 | 0 | 1
  Cholesterol (mg/dl) >1.3 x ULN | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities-urinalysis (Chronic Period)
Description: The number of participants with a laboratory abnormality meeting specified criteria while on study treatment or during lag time are reported here. Baseline is defined as the last measurement prior to receiving study treatment. The list of urinalysis test parameters were as follows:pH, glucose (qual), protein (qual), blood (qual), ketones, nitrites, leukocyte esterase, microscopy, and spot urine albumin/creatinine ratio. The criteria of laboratory abnormality is defined as one of the following conditions was met: 1)associated with accompanying symptoms;2)Test result requires additional diagnostic testing or medical/surgical intervention;3)Test result leads to a change in study dosing (outside of any protocol specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy;4)Test result is considered to be an AE by the investigator or sponsor.
Time Frame: Week 8 to Week 32
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
Number analyzed (Participants) | 35 | 36 | 39 | 10 | 38 | 37 | 39 | 9 | 37
Participants
  pH (scalar) <4.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  pH (scalar) >8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Glucose (No Unit) >=1 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 1
  Ketones (No Unit) >=1 | 4 | 3 | 8 | 2 | 4 | 1 | 3 | 0 | 2
  Urine Protein (No Unit) >=1 | 0 | 1 | 3 | 0 | 1 | 0 | 2 | 0 | 1
  Urine Hemoglobin (No Unit) >=1 | 7 | 4 | 5 | 1 | 7 | 9 | 9 | 0 | 9
  Nitrite (No Unit) >=1 | 2 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 1
  Leukocyte Esterase (No Unit) >=1 | 8 | 13 | 11 | 1 | 14 | 7 | 8 | 1 | 9
  Urine Erythrocytes (/HPF) >=20: number analyzed (Participants) | 22 | 19 | 25 | 6 | 23 | 18 | 25 | 3 | 25
  Urine Erythrocytes (/HPF) >=20 | 1 | 1 | 4 | 1 | 2 | 3 | 5 | 0 | 1
  Urine Leukocytes (/HPF) >=20: number analyzed (Participants) | 25 | 23 | 31 | 9 | 29 | 28 | 29 | 7 | 26
  Urine Leukocytes (/HPF) >=20 | 0 | 2 | 3 | 1 | 3 | 1 | 1 | 0 | 4
  Hyaline Casts (/LPF) >1: number analyzed (Participants) | 7 | 1 | 8 | 3 | 9 | 2 | 6 | 1 | 3
  Hyaline Casts (/LPF) >1 | 5 | 0 | 6 | 2 | 4 | 1 | 2 | 1 | 2
  WBC Casts (/LPF) >1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  WBC Casts (/LPF) >1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bacteria (No Unit) >20: number analyzed (Participants) | 10 | 9 | 10 | 5 | 12 | 9 | 10 | 2 | 12
  Bacteria (No Unit) >20 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Discontinuation Due to AEs (All-causalities) (Induction Period)
Description: as for outcome 2
Time Frame: From Day 1 up to Week 8
Population: The participants who received at least one dose of PF-06651600, PF-06700841, or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Participants
  Participants with AEs | 13 | 23 | 21 | 21 | 19 | 26 | 23
  Participants with SAEs | 0 | 3 | 0 | 3 | 1 | 3 | 1
  Participants discontinued from study due to AEs | 0 | 5 | 0 | 5 | 1 | 2 | 1

11. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Induction Period)
Description: The number of participants with a laboratory abnormality meeting the pre-specified criteria defined in the study protocol while on study treatment or during lag time are reported here. Baseline is defined as the last measurement prior to receiving study treatment. Laboratory data included hematology test, serum chemistry test, C-creative protein and viral surveillance. The criteria of laboratory abnormality is defined as one of the following conditions was met: 1)associated with accompanying symptoms;2)Test result requires additional diagnostic testing or medical/surgical intervention;3)Test result leads to a change in study dosing (outside of any protocol specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy;4)Test result is considered to be an AE by the investigator or sponsor.
Time Frame: From Day 1 up to Week 8
Population: The participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
Participants | 17 | 29 | 28 | 34 | 32 | 31 | 36

12. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities-hematology (Induction Period)
Description: as for outcome 4
Time Frame: From Day 1 up to Week 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Participants
  Hemoglobin (g/dL) <0.8× lower limit of normal (LLN): number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Hemoglobin (g/dL) <0.8× lower limit of normal (LLN) | 3 | 2 | 5 | 9 | 4 | 4 | 5
  Hematocrit (%) <0.8× LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Hematocrit (%) <0.8× LLN | 2 | 0 | 3 | 4 | 1 | 1 | 0
  Erythrocytes (10^6/mm^3) <0.8× LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Erythrocytes (10^6/mm^3) <0.8× LLN | 0 | 0 | 4 | 3 | 1 | 1 | 2
  Reticulocytes (Abs) (10^3/mm^3) <0.5× LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 46 | 47
  Reticulocytes (Abs) (10^3/mm^3) <0.5× LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocytes (Abs) (10^3/mm^3) >1.5× upper limit of normal (ULN): number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 46 | 47
  Reticulocytes (Abs) (10^3/mm^3) >1.5× upper limit of normal (ULN) | 1 | 1 | 2 | 2 | 0 | 0 | 0
  Erythrocytes Mean Corpuscular Volume (10^-15L) <0.9× LLN: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Erythrocytes Mean Corpuscular Volume (10^-15L) <0.9× LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes Mean Corpuscular Volume (10^-15L) >1.1× ULN: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Erythrocytes Mean Corpuscular Volume (10^-15L) >1.1× ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (10^3/mm^3) <0.5× LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Platelets (10^3/mm^3) <0.5× LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (10^3/mm^3) >1.75× ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Platelets (10^3/mm^3) >1.75× ULN | 1 | 0 | 0 | 0 | 2 | 2 | 5
  Reticulocytes/Erythrocytes (%) <0.5× LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 46 | 47
  Reticulocytes/Erythrocytes (%) <0.5× LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocytes/Erythrocytes (%) >1.5× ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 46 | 47
  Reticulocytes/Erythrocytes (%) >1.5× ULN | 1 | 2 | 3 | 3 | 0 | 0 | 2
  Leukocytes (10^3/mm^3) <0.6× LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Leukocytes (10^3/mm^3) <0.6× LLN | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Leukocytes (10^3/mm^3) >1.5× ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Leukocytes (10^3/mm^3) >1.5× ULN | 0 | 3 | 0 | 3 | 2 | 2 | 1
  Lymphocytes (Abs) (10^3/mm^3) <0.8× LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Lymphocytes (Abs) (10^3/mm^3) <0.8× LLN | 3 | 2 | 4 | 11 | 2 | 1 | 2
  Lymphocytes (Abs) (10^3/mm^3) >1.2× ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Lymphocytes (Abs) (10^3/mm^3) >1.2× ULN | 0 | 1 | 0 | 0 | 1 | 1 | 1
  Neutrophils (Abs) (10^3/mm^3) <0.8× LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Neutrophils (Abs) (10^3/mm^3) <0.8× LLN | 1 | 0 | 0 | 0 | 2 | 3 | 2
  Neutrophils (Abs) (10^3/mm^3) >1.2× ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Neutrophils (Abs) (10^3/mm^3) >1.2× ULN | 7 | 13 | 7 | 9 | 7 | 7 | 11
  Basophils (Abs) (10^3/mm^3) >1.2× ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Basophils (Abs) (10^3/mm^3) >1.2× ULN | 0 | 0 | 1 | 0 | 1 | 1 | 0
  Eosinophils (Abs) (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Eosinophils (Abs) (10^3/mm^3) >1.2x ULN | 2 | 3 | 1 | 1 | 1 | 3 | 2
  Monocytes (Abs) (10^3/mm^3) >1.2× ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Monocytes (Abs) (10^3/mm^3) >1.2× ULN | 2 | 2 | 0 | 2 | 1 | 1 | 2
  Activated PTT (second) >1.1× ULN: number analyzed (Participants) | 25 | 48 | 48 | 50 | 48 | 47 | 46
  Activated PTT (second) >1.1× ULN | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PT (second) >1.1× ULN: number analyzed (Participants) | 25 | 48 | 48 | 50 | 48 | 47 | 46
  PT (second) >1.1× ULN | 1 | 2 | 1 | 1 | 0 | 0 | 0
  Prothrombin INR >1.1× ULN: number analyzed (Participants) | 25 | 48 | 48 | 50 | 48 | 47 | 46
  Prothrombin INR >1.1× ULN | 1 | 2 | 1 | 1 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities-clinical Chemistry (Induction Period)
Description: as for outcome 8
Time Frame: From Day 1 up to Week 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Participants
  Bilirubin (mg/dL) >1.5x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Bilirubin (mg/dL) >1.5x ULN | 0 | 1 | 0 | 1 | 2 | 2 | 1
  Direct Bilirubin (mg/dL) >1.5x ULN: number analyzed (Participants) | 2 | 3 | 2 | 5 | 5 | 4 | 2
  Direct Bilirubin (mg/dL) >1.5x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin (mg/dL) >1.5x ULN: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 1
  Indirect Bilirubin (mg/dL) >1.5x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L) >3.0x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  AST (U/L) >3.0x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) >3.0x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  ALT (U/L) >3.0x ULN | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Gamma Glutamyl Transferase (U/L) >3.0x ULN: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 2 | 1
  Gamma Glutamyl Transferase (U/L) >3.0x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L) >3.0x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Alkaline Phosphatase (U/L) >3.0x ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Protein (g/dL) <0.8x LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Protein (g/dL) <0.8x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein (g/dL) >1.2x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Protein (g/dL) >1.2x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) <0.8x LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Albumin (g/dL) <0.8x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) >1.2x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Albumin (g/dL) >1.2x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen (mg/dL) >1.3x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Urea Nitrogen (mg/dL) >1.3x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) >1.3x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 47 | 47 | 47
  Creatinine (mg/dL) >1.3x ULN | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Urate (mg/dL) >1.2x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Urate (mg/dL) >1.2x ULN | 0 | 0 | 1 | 0 | 0 | 0 | 0
  HDL Cholesterol (mg/dL) <0.8x LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  HDL Cholesterol (mg/dL) <0.8x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LDL Cholesterol (mg/dL) >1.2x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  LDL Cholesterol (mg/dL) >1.2x ULN | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Triglycerides (mg/dL) >1.3x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Triglycerides (mg/dL) >1.3x ULN | 1 | 1 | 1 | 3 | 1 | 2 | 5
  Sodium(Meq/L) <0.95x LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Sodium(Meq/L) <0.95x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium(Meq/L) >1.05x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Sodium(Meq/L) >1.05x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (Meq/L) <0.9x LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Potassium (Meq/L) <0.9x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (Meq/L) >1.1x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Potassium (Meq/L) >1.1x ULN | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Chloride (Meq/L) <0.9x LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Chloride (Meq/L) <0.9x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride (Meq/L) >1.1x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Chloride (Meq/L) >1.1x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) <0.9x LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Calcium (mg/dL) <0.9x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) >1.1x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Calcium (mg/dL) >1.1x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) <0.6x LLN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Glucose (mg/dL) <0.6x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) >1.5x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Glucose (mg/dL) >1.5x ULN | 0 | 1 | 2 | 1 | 1 | 0 | 2
  Hemoglobin A1C (%) >1.3x ULN: number analyzed (Participants) | 0 | 2 | 1 | 1 | 0 | 1 | 2
  Hemoglobin A1C (%) >1.3x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CK (U/L) >2.0x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  CK (U/L) >2.0x ULN | 2 | 0 | 2 | 3 | 2 | 3 | 6
  Cholesterol (mg/dl) >1.3x ULN: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Cholesterol (mg/dl) >1.3x ULN | 0 | 0 | 1 | 0 | 0 | 1 | 0

14. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities- Urinalysis (Induction Period)
Description: as for outcome 9
Time Frame: From Day 1 up to Week 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Participants
  pH (scalar) <4.5: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  pH (scalar) <4.5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  pH (scalar) >8: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  pH (scalar) >8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine glucose (no unit) ≥1: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Urine glucose (no unit) ≥1 | 0 | 1 | 4 | 1 | 0 | 1 | 1
  Ketones (no unit) ≥1: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Ketones (no unit) ≥1 | 1 | 4 | 1 | 1 | 7 | 4 | 4
  Urine protein(no unit) ≥1: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Urine protein(no unit) ≥1 | 0 | 2 | 0 | 1 | 1 | 2 | 0
  Urine hemoglobin(no unit) ≥1: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Urine hemoglobin(no unit) ≥1 | 2 | 4 | 4 | 4 | 5 | 8 | 4
  Nitrite (no unit) ≥1: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Nitrite (no unit) ≥1 | 1 | 1 | 2 | 1 | 2 | 0 | 1
  Leukocyte esterase (no unit) ≥1: number analyzed (Participants) | 25 | 49 | 48 | 50 | 48 | 47 | 47
  Leukocyte esterase (no unit) ≥1 | 3 | 11 | 4 | 10 | 7 | 8 | 14
  Urine erythrocytes (/HPF) ≥20: number analyzed (Participants) | 9 | 26 | 19 | 20 | 18 | 26 | 18
  Urine erythrocytes (/HPF) ≥20 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Urine leukocytes (/HPF) ≥20: number analyzed (Participants) | 15 | 33 | 24 | 29 | 31 | 31 | 32
  Urine leukocytes (/HPF) ≥20 | 1 | 2 | 1 | 4 | 3 | 1 | 3
  Granular casts (/LPF) >1: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0 | 0
  Granular casts (/LPF) >1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Hyaline casts (/LPF) >1: number analyzed (Participants) | 3 | 3 | 4 | 4 | 5 | 4 | 2
  Hyaline casts (/LPF) >1 | 3 | 2 | 2 | 4 | 4 | 2 | 1
  WBC casts (/LPF) >1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  WBC casts (/LPF) >1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Bacteria (no unit) >20: number analyzed (Participants) | 5 | 9 | 9 | 9 | 10 | 16 | 11
  Bacteria (no unit) >20 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Abnormal Vital Signs Data (Induction Period)
Description: as for outcome 5
Time Frame: From screening to Week 8
Population: Number of participants evaluated against the criteria during the induction period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 48 | 48 | 49 | 47 | 46 | 45
Participants
  Sitting Systolic Blood Pressure Value <90 mmHg | 0 | 1 | 1 | 0 | 3 | 0 | 0
  Sitting Systolic Blood Pressure Change ≥30 mmHg Increase: number analyzed (Participants) | 21 | 44 | 43 | 41 | 45 | 43 | 44
  Sitting Systolic Blood Pressure Change ≥30 mmHg Increase | 0 | 1 | 3 | 0 | 0 | 0 | 3
  Sitting Systolic Blood Pressure Change ≥30 mmHg Decrease | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Sitting Diastolic Blood Pressure Value <50 mmHg | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Sitting Diastolic Blood Pressure Change ≥20 mmHg Increase | 0 | 2 | 3 | 0 | 2 | 1 | 5
  Sitting Diastolic Blood Pressure Change ≥20 mmHg Decrease | 0 | 4 | 4 | 2 | 2 | 1 | 2
  Sitting Pulse Rate Value <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting Pulse Rate Value >120 bpm | 0 | 1 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings (Induction Period)
Description: The number of participants with abnormal ECG findings during the induction period (from Day 1 to Week 8) are reported below. The criteria of test abnormality is defined as one of the following conditions was met: 1)associated with accompanying symptoms;2)Test result requires additional diagnostic testing or medical/surgical intervention;3)Test result leads to a change in study dosing (outside of any protocol specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy;4)Test result is considered to be an AE by the investigator or sponsor.
Time Frame: From screening to Week 8
Population: Number of Participants Analyzed: the participants who received at least one dose of PF-06651600, PF-06700841, or placebo. Number Analyzed: the participants evaluated at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Participants
  abnormal, not clinical significant (at screening) | 2 | 8 | 6 | 4 | 9 | 10 | 8
  abnormal, clinical significant (at screening) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  abnormal, not clinical significant (at Week 8): number analyzed (Participants) | 20 | 42 | 42 | 40 | 44 | 42 | 43
  abnormal, not clinical significant (at Week 8) | 2 | 7 | 8 | 4 | 5 | 4 | 3
  abnormal, clinical significant (at Week 8): number analyzed (Participants) | 20 | 42 | 42 | 40 | 44 | 42 | 43
  abnormal, clinical significant (at Week 8) | 0 | 0 | 0 | 1 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Serious Infections (Induction Period)
Description: Serious infections was defined as any infection (for example, viral, bacterial, and fungal) requiring hospitalization or parenteral antimicrobials including Listeria encephalitis, Pneumonia, Viral infection.
Time Frame: From Day 1 up to Week 8
Population: The participants who received at least one dose of PF-06651600, PF-06700841, or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Participants
  Listeria encephalitis | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Pneumonia | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Viral infection | 0 | 1 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants Achieving Remission Based on Total Mayo Score at Week 8 (Induction Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity. Clinical remission was defined as total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0.
Time Frame: Week 8
Population: The ITT analysis set which included all randomized participants who received at least 1 dose of investigational product or placebo.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants | 0 [0.0 to 11.0] | 9.8 [4.8 to 19.1] | 28.6 [19.0 to 40.4] | 34.0 [24.0 to 45.4] | 8.3 [3.7 to 16.8] | 23.4 [14.8 to 34.5] | 23.4 [14.8 to 34.5]
Statistical Analysis 1: Comparison: Placebo (Induction) vs PF-06651600 20 mg (Induction); Test type: Superiority; p = 0.0626, Chan and Zhang method; Mean Difference (Final Values) = 9.8, 90% CI 2-sided [-1.0 to 19.5]
Statistical Analysis 2: Comparison: Placebo (Induction) vs PF-06651600 70 mg (Induction); Test type: Superiority; p = 0.0027, Chan and Zhang method; Mean Difference (Final Values) = 28.6, 90% CI 2-sided [13.9 to 41.0]
Statistical Analysis 3: Comparison: Placebo (Induction) vs PF-06651600 200 mg (Induction); Test type: Superiority; p = 0.0010, Chan and Zhang Method; Mean Difference (Final Values) = 34.0, 90% CI 2-sided [20.2 to 46.5]
Statistical Analysis 4: Comparison: Placebo (Induction) vs PF-06700841 10 mg (Induction); Test type: Superiority; p = 0.0774, Chan and Zhang method; Mean Difference (Final Values) = 8.3, 90% CI 2-sided [-4.0 to 18.1]
Statistical Analysis 5: Comparison: Placebo (Induction) vs PF-06700841 30 mg (Induction); Test type: Superiority; p = 0.0055, Chan and Zhang method; Mean Difference (Final Values) = 23.4, 90% CI 2-sided [8.2 to 35.8]
Statistical Analysis 6: Comparison: Placebo (Induction) vs PF-06700841 60 mg (Induction); Test type: Superiority; p = 0.0055, Chan and Zhang method; Mean Difference (Final Values) = 23.4, 90% CI 2-sided [8.2 to 35.8]

19. Secondary Outcome: Percentage of Participants Achieving Improvement in Endoscopic Appearance Based on Total Mayo Score at Week 8 (Induction Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity. Improvement in endoscopic subscore appearance was defined at Mayo endoscopic subscore of ≤1.
Time Frame: Week 8
Population: as for outcome 18
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants | 0 [0.0 to 11.0] | 21.6 [13.5 to 33.1] | 34.7 [24.4 to 46.4] | 42.0 [30.3 to 54.6] | 20.8 [11.8 to 31.5] | 31.9 [20.8 to 44.4] | 29.8 [19.9 to 42.3]
Statistical Analysis 1: Comparison: Placebo (Induction) vs PF-06651600 20 mg (Induction); Test type: Superiority; p = 0.0111, Chan and Zhang method; Mean Difference (Final Values) = 21.6, 90% CI 2-sided [5.6 to 33.2]
Statistical Analysis 2: Comparison: Placebo (Induction) vs PF-06651600 70 mg (Induction); Test type: Superiority; p = 0.0006, Chan and Zhang method; Mean Difference (Final Values) = 34.7, 90% CI 2-sided [20.2 to 47.4]
Statistical Analysis 3: Comparison: Placebo (Induction) vs PF-06651600 200 mg (Induction); Test type: Superiority; p = 0.0001, Chan and Zhang Method; Mean Difference (Final Values) = 42.0, 90% CI 2-sided [29.5 to 54.6]
Statistical Analysis 4: Comparison: Placebo (Induction) vs PF-06700841 10 mg (Induction); Test type: Superiority; p = 0.0101, Chan and Zhang method; Mean Difference (Final Values) = 20.8, 90% CI 2-sided [5.6 to 33.0]
Statistical Analysis 5: Comparison: Placebo (Induction) vs PF-06700841 30 mg (Induction); Test type: Superiority; p = 0.0014, Chan and Zhang method; Mean Difference (Final Values) = 31.9, 90% CI 2-sided [17.0 to 44.8]
Statistical Analysis 6: Comparison: Placebo (Induction) vs PF-06700841 60 mg (Induction); Test type: Superiority; p = 0.0015, Chan and Zhang method; Mean Difference (Final Values) = 29.8, 90% CI 2-sided [17.0 to 42.6]

20. Secondary Outcome: Percentage of Participants Achieving Clinical Response Based on Total Mayo Score at Week 8 (Induction Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity. Clinical response was defined as decrease from baseline in total Mayo score of at least 3 points and at least 30%, with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or absolute subscore for rectal bleeding of 0 or 1.
Time Frame: Week 8
Population: as for outcome 18
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants | 24.0 [11.0 to 41.7] | 41.2 [29.9 to 53.6] | 69.4 [57.6 to 80.1] | 68.0 [56.6 to 78.8] | 41.7 [29.6 to 54.5] | 53.2 [40.3 to 65.5] | 61.7 [48.7 to 72.9]
Statistical Analysis 1: Comparison: Placebo (Induction) vs PF-06651600 20 mg (Induction); Test type: Superiority; p = 0.0788, Chan and Zhang method; Mean Difference (Final Values) = 17.2, 90% CI 2-sided [-3.4 to 34.4]
Statistical Analysis 2: Comparison: Placebo (Induction) vs PF-06651600 70 mg (Induction); Test type: Superiority; p = 0.0002, Chan and Zhang method; Mean Difference (Final Values) = 45.4, 90% CI 2-sided [23.6 to 62.1]
Statistical Analysis 3: Comparison: Placebo (Induction) vs PF-06651600 200 mg (Induction); Test type: Superiority; p = 0.0003, Chan and Zhang Method; Mean Difference (Final Values) = 44.0, 90% CI 2-sided [23.5 to 60.5]
Statistical Analysis 4: Comparison: Placebo (Induction) vs PF-06700841 10 mg (Induction); Test type: Superiority; p = 0.0773, Chan and Zhang method; Mean Difference (Final Values) = 17.7, 90% CI 2-sided [-4.0 to 35.1]
Statistical Analysis 5: Comparison: Placebo (Induction) vs PF-06700841 30 mg (Induction); Test type: Superiority; p = 0.0136, Chan and Zhang method; Mean Difference (Final Values) = 29.2, 90% CI 2-sided [5.6 to 47.0]
Statistical Analysis 6: Comparison: Placebo (Induction) vs PF-06700841 60 mg (Induction); Test type: Superiority; p = 0.0015, Chan and Zhang method; Mean Difference (Final Values) = 37.7, 90% CI 2-sided [13.9 to 54.7]

21. Secondary Outcome: Percentage of Participants Achieving Endoscopic Remission Based on Total Mayo Score at Week 8 (Induction Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity. Endoscopic remission was defined as endoscopic subscore of 0.
Time Frame: Week 8
Population: as for outcome 18
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants | 0 [0.0 to 11.0] | 3.9 [1.0 to 11.0] | 8.2 [3.6 to 16.5] | 12.0 [5.4 to 21.2] | 2.1 [0.2 to 8.6] | 17.0 [8.8 to 28.3] | 8.5 [3.8 to 17.2]
Statistical Analysis 1: Comparison: Placebo (Induction) vs PF-06651600 20 mg (Induction); Test type: Superiority; p = 0.2259, Chan and Zhang method; Mean Difference (Final Values) = 3.9, 90% CI 2-sided [-6.5 to 11.8]
Statistical Analysis 2: Comparison: Placebo (Induction) vs PF-06651600 70 mg (Induction); Test type: Superiority; p = 0.0820, Chan and Zhang method; Mean Difference (Final Values) = 8.2, 90% CI 2-sided [-3.8 to 17.7]
Statistical Analysis 3: Comparison: Placebo (Induction) vs PF-06651600 200 mg (Induction); Test type: Superiority; p = 0.0649, Chan and Zhang Method; Mean Difference (Final Values) = 12.0, 90% CI 2-sided [-0.7 to 22.3]
Statistical Analysis 4: Comparison: Placebo (Induction) vs PF-06700841 10 mg (Induction); Test type: Superiority; p = 0.3777, Chan and Zhang method; Mean Difference (Final Values) = 2.1, 90% CI 2-sided [-8.6 to 9.7]
Statistical Analysis 5: Comparison: Placebo (Induction) vs PF-06700841 30 mg (Induction); Test type: Superiority; p = 0.0212, Chan and Zhang method; Mean Difference (Final Values) = 17.0, 90% CI 2-sided [2.9 to 28.6]
Statistical Analysis 6: Comparison: Placebo (Induction) vs PF-06700841 60 mg (Induction); Test type: Superiority; p = 0.0742, Chan and Zhang method; Mean Difference (Final Values) = 8.5, 90% CI 2-sided [-4.2 to 18.4]

22. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission Based on Total Mayo Score at Week 8 (Induction Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity. Symptomatic remission was defined as total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point, and both rectal bleeding and stool frequency subscores of 0.
Time Frame: Week 8
Population: as for outcome 18
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants | 0 [0.0 to 11.0] | 7.8 [3.5 to 15.9] | 16.3 [8.4 to 27.1] | 26.0 [16.2 to 37.6] | 6.3 [2.3 to 15.1] | 14.9 [8.0 to 25.1] | 14.9 [8.0 to 25.1]
Statistical Analysis 1: Comparison: Placebo (Induction) vs PF-06651600 20 mg (Induction); Test type: Superiority; p = 0.0872, Chan and Zhang method; Mean Difference (Final Values) = 7.8, 90% CI 2-sided [-3.4 to 17.1]
Statistical Analysis 2: Comparison: Placebo (Induction) vs PF-06651600 70 mg (Induction); Test type: Superiority; p = 0.0254, Chan and Zhang method; Mean Difference (Final Values) = 16.3, 90% CI 2-sided [3.0 to 27.5]
Statistical Analysis 3: Comparison: Placebo (Induction) vs PF-06651600 200 mg (Induction); Test type: Superiority; p = 0.0034, Chan and Zhang Method; Mean Difference (Final Values) = 26.0, 90% CI 2-sided [11.0 to 38.1]
Statistical Analysis 4: Comparison: Placebo (Induction) vs PF-06700841 10 mg (Induction); Test type: Superiority; p = 0.1565, Chan and Zhang method; Mean Difference (Final Values) = 6.3, 90% CI 2-sided [-4.5 to 15.4]
Statistical Analysis 5: Comparison: Placebo (Induction) vs PF-06700841 30 mg (Induction); Test type: Superiority; p = 0.0288, Chan and Zhang method; Mean Difference (Final Values) = 14.9, 90% CI 2-sided [1.7 to 26.2]
Statistical Analysis 6: Comparison: Placebo (Induction) vs PF-06700841 60 mg (Induction); Test type: Superiority; p = 0.0288, Chan and Zhang method; Mean Difference (Final Values) = 14.9, 90% CI 2-sided [1.7 to 26.2]

23. Secondary Outcome: Percentage of Participants Achieving Deep Remission Based on Total Mayo Score at Week 8 (Induction Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity. Deep remission was defined as total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a zero on both endoscopic and rectal bleeding subscore.
Time Frame: Week 8
Population: as for outcome 18
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants | 0 [0.0 to 11.0] | 3.9 [1.0 to 11.0] | 8.2 [3.6 to 16.5] | 12.0 [5.4 to 21.2] | 0 [0.0 to 5.6] | 14.9 [8.0 to 25.1] | 6.4 [2.4 to 15.4]
Statistical Analysis 1: Comparison: Placebo (Induction) vs PF-06651600 20 mg (Induction); Test type: Superiority; p = 0.2259, Chan and Zhang method; Mean Difference (Final Values) = 3.9, 90% CI 2-sided [-6.5 to 11.8]
Statistical Analysis 2: Comparison: Placebo (Induction) vs PF-06651600 70 mg (Induction); Test type: Superiority; p = 0.0820, Chan and Zhang method; Mean Difference (Final Values) = 8.2, 90% CI 2-sided [-3.8 to 17.7]
Statistical Analysis 3: Comparison: Placebo (Induction) vs PF-06651600 200 mg (Induction); Test type: Superiority; p = 0.0649, Chan and Zhang Method; Mean Difference (Final Values) = 12.0, 90% CI 2-sided [-0.7 to 22.3]
Statistical Analysis 4: Comparison: Placebo (Induction) vs PF-06700841 10 mg (Induction); Test type: Superiority; p = 1.0000, Chan and Zhang method; Mean Difference (Final Values) = 0.0, 90% CI 2-sided [-11.3 to 6.1]
Statistical Analysis 5: Comparison: Placebo (Induction) vs PF-06700841 30 mg (Induction); Test type: Superiority; p = 0.0288, Chan and Zhang method; Mean Difference (Final Values) = 14.9, 90% CI 2-sided [1.7 to 26.2]
Statistical Analysis 6: Comparison: Placebo (Induction) vs PF-06700841 60 mg (Induction); Test type: Superiority; p = 0.1593, Chan and Zhang method; Mean Difference (Final Values) = 6.4, 90% CI 2-sided [-4.4 to 15.7]

24. Secondary Outcome: Partial Mayo Score and Change From Baseline at Weeks 2, 4 and 8 (Induction Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity. The partial Mayo score does not incorporate the endoscopy score and the partial Mayo score ranges from 0 to 9.
Time Frame: Baseline, Weeks 2, 4 and 8
Population: Number of Participants Analyzed: ITT analysis set which included all participants who were randomized to the study and received at least one dose of the randomized investigational drug. Number Analyzed: the participants in the ITT analysis set who had partial Mayo score at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Units on a scale
  Week 2: number analyzed (Participants) | 24 | 49 | 48 | 46 | 45 | 45 | 45
  Week 2 | -0.66 (0.37) | -1.65 (0.26) | -2.56 (0.26) | -3.19 (0.27) | -1.6 (0.27) | -1.64 (0.27) | -2.45 (0.27)
  Week 4: number analyzed (Participants) | 23 | 48 | 46 | 42 | 47 | 44 | 44
  Week 4 | -1.64 (0.42) | -2.24 (0.29) | -3.29 (0.30) | -4.24 (0.31) | -2.31 (0.30) | -2.06 (0.30) | -2.95 (0.30)
  Week 8: number analyzed (Participants) | 22 | 45 | 46 | 40 | 45 | 44 | 44
  Week 8 | -1.15 (0.43) | -2.54 (0.30) | -4.06 (0.30) | -4.69 (0.32) | -2.51 (0.30) | -2.71 (0.31) | -3.47 (0.31)

25. Secondary Outcome: Change From Baseline in Total Mayo Score at Week 8 (Induction Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Units on a scale | -1.14 [-2.06 to -0.22] | -3.17 [-3.83 to -2.51] | -5.02 [-5.68 to -4.36] | -5.74 [-6.43 to -5.06] | -2.93 [-3.58 to -2.29] | -3.42 [-4.08 to -2.76] | -4.35 [-5.00 to -3.69]

26. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Domain Score and Total Score at Weeks 4 and 8 (Induction Period)
Description: IBDQ is a psychometrically validated patient reported outcome (PRO) instrument for measuring the disease specific quality of life in participants with inflammatory bowel disease (IBD). The IBDQ is comprised of 32 items, which are grouped into 4 dimensions: bowel function, emotional status, systemic symptoms and social function. The 4 domains are scored as follows: Bowel symptoms: 10 to 70; Systemic symptoms: 5 to 35.; Emotional function: 12 to 84; Social function: 5 to 35. The total IBDQ score ranges from 32 to 224. For the total score and each domain, a higher score indicates better quality of life.
Time Frame: Week 4 and Week 8
Population: Number of Participants Analyzed: ITT analysis set includes all participants who were randomized to the study and received at least one dose of the randomized investigational drug. Number Analyzed: the participants evaluated for IBDQ at each specified time point.
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Units on a scale
  Baseline (Bowel Systems Domain score): number analyzed (Participants) | 25 | 51 | 49 | 49 | 47 | 47 | 47
  Baseline (Bowel Systems Domain score) | 35.80 [32.48 to 39.12] | 34.29 [31.74 to 36.85] | 33.71 [31.41 to 36.01] | 34.84 [32.66 to 37.01] | 34.17 [32.13 to 36.21] | 32.38 [29.99 to 34.77] | 33.38 [31.36 to 35.40]
  Week 4 (Bowel Systems Domain score): number analyzed (Participants) | 23 | 46 | 47 | 44 | 46 | 44 | 44
  Week 4 (Bowel Systems Domain score) | 44.87 [40.65 to 49.09] | 46.98 [44.05 to 49.91] | 51.00 [48.45 to 53.55] | 53.80 [50.83 to 56.76] | 44.93 [42.00 to 47.86] | 46.84 [43.56 to 50.12] | 50.64 [47.66 to 53.61]
  Week 8 (Bowel Systems Domain score): number analyzed (Participants) | 22 | 47 | 45 | 41 | 45 | 43 | 44
  Week 8 (Bowel Systems Domain score) | 44.68 [41.37 to 47.99] | 47.96 [44.68 to 51.23] | 54.27 [51.38 to 57.16] | 55.95 [53.40 to 58.50] | 46.87 [43.46 to 50.27] | 50.12 [47.12 to 53.11] | 53.45 [50.53 to 56.38]
  Baseline (Emotion Health Domain score): number analyzed (Participants) | 25 | 51 | 49 | 49 | 47 | 47 | 47
  Baseline (Emotion Health Domain score) | 43.76 [38.81 to 48.71] | 42.76 [39.37 to 46.16] | 42.90 [39.56 to 46.24] | 41.39 [37.88 to 44.90] | 42.40 [39.15 to 45.65] | 38.74 [35.59 to 41.90] | 41.43 [38.56 to 44.29]
  Week 4(Emotion Health Domain score): number analyzed (Participants) | 23 | 46 | 47 | 44 | 46 | 44 | 44
  Week 4(Emotion Health Domain score) | 54.74 [49.67 to 59.81] | 53.65 [49.92 to 57.39] | 59.89 [56.83 to 62.96] | 61.11 [57.54 to 64.68] | 52.43 [48.26 to 56.61] | 52.77 [48.99 to 56.55] | 57.86 [54.06 to 61.67]
  Week 8(Emotion Health Domain score): number analyzed (Participants) | 22 | 47 | 45 | 41 | 45 | 43 | 44
  Week 8(Emotion Health Domain score) | 52.50 [47.61 to 57.39] | 54.23 [50.29 to 58.17] | 62.73 [59.30 to 66.17] | 63.12 [59.28 to 66.96] | 54.44 [50.02 to 58.87] | 56.86 [53.34 to 60.38] | 60.89 [57.09 to 64.69]
  Baseline (Systemic Systems Domain score): number analyzed (Participants) | 25 | 51 | 49 | 49 | 47 | 47 | 47
  Baseline (Systemic Systems Domain score) | 16.56 [14.83 to 18.29] | 16.12 [14.74 to 17.50] | 15.98 [14.67 to 17.29] | 15.41 [14.14 to 16.68] | 16.30 [14.93 to 17.67] | 15.21 [14.06 to 16.36] | 16.72 [15.40 to 18.05]
  Week 4(Systemic Systems Domain score): number analyzed (Participants) | 23 | 46 | 47 | 44 | 46 | 44 | 44
  Week 4(Systemic Systems Domain score) | 20.87 [18.56 to 23.18] | 21.70 [20.34 to 23.05] | 23.74 [22.44 to 25.05] | 23.66 [22.08 to 25.23] | 20.70 [19.03 to 22.36] | 20.77 [19.24 to 22.30] | 23.61 [21.89 to 25.34]
  Week 8(Systemic Systems Domain score): number analyzed (Participants) | 22 | 47 | 45 | 41 | 45 | 43 | 44
  Week 8(Systemic Systems Domain score) | 20.82 [19.11 to 22.53] | 21.85 [20.20 to 23.50] | 24.40 [22.91 to 25.89] | 25.51 [24.17 to 26.86] | 21.40 [19.56 to 23.24] | 23.07 [21.50 to 24.64] | 24.48 [22.72 to 26.24]
  Baseline (Social Function Domain score): number analyzed (Participants) | 25 | 51 | 49 | 49 | 47 | 47 | 47
  Baseline (Social Function Domain score) | 16.88 [14.41 to 19.35] | 17.25 [15.43 to 19.08] | 16.59 [14.70 to 18.48] | 17.31 [15.73 to 18.88] | 17.30 [15.69 to 18.91] | 14.91 [13.28 to 16.55] | 16.64 [15.06 to 18.22]
  Week 4 (Social Function Domain score): number analyzed (Participants) | 23 | 46 | 47 | 44 | 46 | 44 | 44
  Week 4 (Social Function Domain score) | 22.57 [19.80 to 25.33] | 22.41 [20.57 to 24.25] | 26.21 [24.73 to 27.70] | 28.20 [26.42 to 29.99] | 22.83 [20.78 to 24.87] | 23.02 [20.82 to 25.23] | 24.86 [22.55 to 27.17]
  Week 8 (Social Function Domain score): number analyzed (Participants) | 22 | 47 | 45 | 41 | 45 | 43 | 44
  Week 8 (Social Function Domain score) | 21.91 [19.27 to 24.55] | 23.45 [21.45 to 25.44] | 27.02 [25.06 to 28.99] | 29.80 [28.14 to 31.47] | 24.36 [22.11 to 26.60] | 25.12 [22.88 to 27.35] | 26.57 [24.50 to 28.63]
  Baseline (Total IBDQ score): number analyzed (Participants) | 25 | 51 | 49 | 49 | 47 | 47 | 47
  Baseline (Total IBDQ score) | 113.00 [101.49 to 124.51] | 110.43 [101.85 to 119.01] | 109.18 [101.30 to 117.07] | 108.94 [101.20 to 116.68] | 110.17 [102.94 to 117.40] | 101.26 [93.85 to 108.66] | 108.17 [101.13 to 115.21]
  Week 4 (Total IBDQ score): number analyzed (Participants) | 23 | 46 | 47 | 44 | 46 | 44 | 44
  Week 4 (Total IBDQ score) | 143.04 [129.90 to 156.19] | 144.74 [135.60 to 153.88] | 160.85 [153.50 to 168.20] | 166.77 [157.55 to 176.00] | 140.89 [130.88 to 150.90] | 143.41 [133.62 to 153.20] | 156.98 [146.69 to 167.27]
  Week 8 (Total IBDQ score): number analyzed (Participants) | 22 | 47 | 45 | 41 | 45 | 43 | 44
  Week 8 (Total IBDQ score) | 139.91 [128.72 to 151.10] | 147.49 [137.17 to 157.80] | 168.42 [159.53 to 177.31] | 174.39 [165.67 to 183.11] | 147.07 [135.79 to 158.35] | 155.16 [145.67 to 164.65] | 165.39 [155.29 to 175.49]

27. Secondary Outcome: Change From Baseline in IBDQ Total Score at Weeks 4 and 8 (Induction Period)
Description: IBDQ is a psychometrically validated PRO instrument for measuring the disease specific quality of life in participants with IBD. The IBDQ is comprised of 32 items, which are grouped into 4 dimensions: bowel function, emotional status, systemic symptoms and social function. The 4 domains are scored as follows: Bowel symptoms: 10 to 70; Systemic symptoms: 5 to 35.; Emotional function: 12 to 84; Social function: 5 to 35. The total IBDQ score ranges from 32 to 224. For the total score and each domain, a higher score indicates better quality of life. Baseline value is defined as the last non-missing measurement collected prior to or on Day 1.
Time Frame: Baseline, Weeks 4 and 8
Population: Number of Participants Analyzed: ITT analysis set includes all participants who were randomized to the study and received at least one dose of the randomized investigational drug. Number Analyzed: The participants with non-missing data in the intent-to-treat analysis set at each specified visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Units on a scale
  Week 4: number analyzed (Participants) | 23 | 46 | 47 | 43 | 45 | 44 | 44
  Week 4 | 30.30 (6.51) | 33.71 (4.60) | 51.12 (4.61) | 57.01 (4.78) | 28.45 (4.68) | 37.94 (4.72) | 49.79 (4.73)
  Week 8: number analyzed (Participants) | 22 | 47 | 45 | 40 | 44 | 43 | 44
  Week 8 | 24.23 (7.40) | 37.91 (5.15) | 59.20 (5.23) | 62.17 (5.47) | 36.60 (5.29) | 48.81 (5.33) | 56.39 (5.33)

28. Secondary Outcome: Percentage of Participants With IBDQ Total Score Greater Than or Equal to 170 at Weeks 4 and 8 (Induction Period)
Description: IBDQ is a psychometrically validated PRO instrument for measuring the disease specific quality of life in participants with IBD. The IBDQ is comprised of 32 items, which are grouped into 4 dimensions: bowel function, emotional status, systemic symptoms and social function. The 4 domains are scored as follows: Bowel symptoms: 10 to 70; Systemic symptoms: 5 to 35.; Emotional function: 12 to 84; Social function: 5 to 35. The total IBDQ score ranges from 32 to 224. For the total score and each domain, a higher score indicates better quality of life.
Time Frame: Week 4 and Week 8
Population: Number of Participants Analyzed: ITT analysis set includes all participants who were randomized to the study and received at least one dose of the randomized investigational drug. Number Analyzed: ITT analysis set which included all participants who were randomized to the study and received at least one dose of the randomized investigational drug, with non-responder imputation of missing data (treating the missing data as non-responders).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants
  Week 4 | 24.0 [11.0 to 41.7] | 21.6 [13.5 to 33.1] | 40.8 [28.9 to 53.6] | 46.0 [34.2 to 58.5] | 27.1 [16.8 to 39.4] | 27.7 [17.2 to 40.3] | 38.3 [27.1 to 51.3]
  Week 8: number analyzed (Participants) | 25 | 51 | 49 | 40 | 48 | 47 | 47
  Week 8 | 20.0 [10.1 to 36.2] | 29.4 [19.1 to 40.6] | 57.1 [44.4 to 69.2] | 44.0 [33.0 to 56.6] | 31.3 [20.4 to 43.4] | 40.4 [28.3 to 53.5] | 51.1 [38.9 to 62.8]

29. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 16 Points Increase in IBDQ Total Score From Baseline at Weeks 4 and 8 (Induction Period)
Description: as for outcome 28
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 28
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants
  Week 4 | 48.0 [30.7 to 64.0] | 60.8 [48.4 to 72.3] | 83.7 [72.9 to 91.6] | 80.0 [69.7 to 88.7] | 64.6 [52.5 to 75.3] | 78.7 [67.8 to 88.0] | 72.3 [59.7 to 82.8]
  Week 8 | 56.0 [38.9 to 73.0] | 54.9 [42.5 to 66.9] | 79.6 [69.2 to 88.5] | 70.0 [58.5 to 80.5] | 62.5 [50.0 to 73.6] | 80.9 [69.7 to 88.8] | 78.7 [67.8 to 88.0]

30. Secondary Outcome: Percentage of Participants With Improvement in IBDQ Bowel Symptom Domain at Weeks 4 and 8 (Induction Period)
Description: IBDQ is a psychometrically validated PRO instrument for measuring the disease specific quality of life in participants with IBD. The IBDQ is comprised of 32 items, which are grouped into 4 dimensions: bowel function, emotional status, systemic symptoms and social function. The 4 domains are scored as follows: Bowel symptoms: 10 to 70; Systemic symptoms: 5 to 35.; Emotional function: 12 to 84; Social function: 5 to 35. The total IBDQ score ranges from 32 to 224. For the total score and each domain, a higher score indicates better quality of life. The improvement in IBDQ bowel symptom domain was defined as an increase of ≥1.2 points from baseline in average score among bowel symptoms domain (items 1, 5, 9, 13, 17, 20, 22, 24, 26, 29).
Time Frame: Week 4 and Week 8
Population: as for outcome 28
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Percentage of participants
  Week 4 | 20.0 [10.1 to 36.2] | 51.0 [38.7 to 63.2] | 65.3 [53.6 to 75.6] | 64.0 [42.6 to 75.1] | 37.5 [26.4 to 50.0] | 53.2 [40.3 to 65.5] | 57.5 [44.4 to 69.7]
  Week 8 | 24.0 [11.0 to 41.7] | 47.1 [35.0 to 59.4] | 69.4 [57.6 to 80.1] | 62.0 [50.0 to 73.5] | 50.0 [37.6 to 62.4] | 63.8 [51.3 to 74.9] | 66.0 [53.5 to 77.3]

31. Secondary Outcome: Change From Baseline in Short Form 36 Version 2 (SF-36v2) Acute Mental Component Summary (MCS) Score and Physical Component Summary (PCS) Score at Weeks 4 and 8 (Induction Period)
Description: The SF-36 version 2 (Acute version) is a 36-item generic health status measure. It measures 8 general health concepts or domains: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), and Mental Health (MH). These 8 domains can also be summarized as physical and mental component scores. The summary component scores, Physical Component Summary (PCS) and Mental Component Summary (MCS), are based on a normalized sum of the 8 scale scores PF, RP, BP, GH, VT, SF, RE, and MH . All domains and summary components are scored such that a higher score indicates a higher functioning or health level. The minimum and maximum scores of the PCS Score are 6.1 and 79.7, respectively. The minimum and maximum scores of the MCS Score are -3.8 and 78.7, respectively.
Time Frame: Week 4 and Week 8
Population: Number of Participants Analyzed: ITT analysis set includes all participants who were randomized to the study and received at least one dose of the randomized investigational drug. Number Analyzed: Number of participants with non-missing data in the ITT analysis set at each specified visit.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Units on a scale
  Week 4 (PCS): number analyzed (Participants) | 23 | 46 | 47 | 43 | 46 | 44 | 44
  Week 4 (PCS) | 4.69 [2.59 to 6.80] | 5.90 [4.41 to 7.39] | 6.36 [4.88 to 7.85] | 9.21 [7.67 to 10.76] | 5.67 [4.16 to 7.19] | 5.85 [4.31 to 7.38] | 6.40 [4.87 to 7.93]
  Week 8 (PCS): number analyzed (Participants) | 22 | 47 | 45 | 40 | 44 | 43 | 44
  Week 8 (PCS) | 5.37 [2.96 to 7.77] | 5.85 [4.19 to 7.52] | 8.66 [6.97 to 10.35] | 10.86 [9.08 to 12.64] | 6.29 [4.57 to 8.02] | 8.21 [6.47 to 9.95] | 8.55 [6.83 to 10.27]
  Week 4(MCS): number analyzed (Participants) | 23 | 46 | 47 | 43 | 46 | 44 | 44
  Week 4(MCS) | 7.83 [4.59 to 11.06] | 4.95 [2.67 to 7.23] | 7.79 [5.50 to 10.07] | 8.81 [6.43 to 11.18] | 2.44 [0.13 to 4.74] | 7.46 [5.11 to 9.82] | 9.28 [6.93 to 11.62]
  Week 8(MCS): number analyzed (Participants) | 22 | 47 | 45 | 40 | 44 | 43 | 44
  Week 8(MCS) | 4.24 [0.69 to 7.78] | 5.18 [2.72 to 7.64] | 9.72 [7.22 to 12.22] | 9.41 [6.79 to 12.03] | 5.22 [2.70 to 7.75] | 8.04 [5.48 to 10.61] | 10.01 [7.47 to 12.55]

32. Secondary Outcome: Change From Baseline in Euro Quality of Life Questionnaire 5 Dimensions 3 Levels (EQ-5D 3L) Utility Score and EQ-5D Visual Analog Scale (VAS) at Weeks 4 and 8 (Induction Period)
Description: For EQ-5D 3L, participant rated questionnaire to assess generic health status in two parts: single utility score and visual analog scale. For utility score, participants rated their current health state on 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression with each dimension having three levels of function: 1 indicates no problem; 2 indicates some problem; 3 indicates extreme problem. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score was transformed and results in a total score range of 0.05 to 1.00; higher scores indicating a better health state. The EQ-5D VAS records the respondent's self rated health on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Week 4 and Week 8
Population: as for outcome 31
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction)
Number analyzed (Participants) | 25 | 51 | 49 | 50 | 48 | 47 | 47
Units on a scale
  EQ-5D 3L Utility Score (Week 4): number analyzed (Participants) | 23 | 46 | 47 | 43 | 46 | 44 | 44
  EQ-5D 3L Utility Score (Week 4) | 0.11 [0.06 to 0.16] | 0.07 [0.04 to 0.11] | 0.12 [0.09 to 0.15] | 0.13 [0.10 to 0.17] | 0.07 [0.03 to 0.10] | 0.11 [0.08 to 0.14] | 0.12 [0.09 to 0.15]
  EQ-5D 3L Utility Score (Week 8): number analyzed (Participants) | 22 | 47 | 45 | 40 | 44 | 43 | 44
  EQ-5D 3L Utility Score (Week 8) | 0.08 [0.03 to 0.13] | 0.08 [0.05 to 0.12] | 0.15 [0.11 to 0.18] | 0.15 [0.12 to 0.19] | 0.09 [0.05 to 0.13] | 0.13 [0.10 to 0.17] | 0.14 [0.11 to 0.18]
  EQ-5D VAS Score (Week 4): number analyzed (Participants) | 23 | 46 | 47 | 43 | 46 | 44 | 44
  EQ-5D VAS Score (Week 4) | 8.41 [2.18 to 14.63] | 13.60 [9.20 to 18.00] | 16.35 [11.96 to 20.74] | 17.45 [12.88 to 22.02] | 10.48 [6.04 to 14.92] | 12.24 [7.72 to 16.77] | 14.44 [9.90 to 18.97]
  EQ-5D VAS Score (Week 8): number analyzed (Participants) | 22 | 47 | 45 | 40 | 44 | 43 | 44
  EQ-5D VAS Score (Week 8) | 13.17 [6.48 to 19.85] | 13.11 [8.48 to 17.74] | 18.88 [14.17 to 23.60] | 22.54 [17.60 to 27.49] | 10.35 [5.58 to 15.12] | 17.11 [12.28 to 21.94] | 20.01 [15.21 to 24.81]

33. Secondary Outcome: Total Mayo Score at Week 32 (Chronic Period)
Description: as for outcome 25
Time Frame: Week 32
Population: The participants with non-missing data at Week 32 in the modified intent-to-treat (MITT) analysis set which included all participants who were randomized to the study and received at least one dose of the randomized investigational drug, but were not randomized to placebo treatment during chronic period.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 200 mg -> PF-06651600 50 mg | Placebo -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg
Number analyzed (Participants) | 10 | 39 | 36 | 35 | 9 | 39 | 38 | 37
Units on a scale | 4.13 [2.82 to 5.44] | 3.47 [2.75 to 4.19] | 3.46 [2.77 to 4.16] | 2.89 [2.18 to 3.60] | 4.62 [2.62 to 6.61] | 3.81 [2.94 to 4.68] | 3.63 [2.67 to 4.59] | 3.86 [2.98 to 4.75]

34. Secondary Outcome: Percentage of Participants Achieving Remission Based on Total Mayo Score at Week 32 (Chronic Period)
Description: as for outcome 18
Time Frame: Week 32
Population: MITT analysis set that included all participants who were randomized to the study and received at least one dose of the randomized investigational drug, but were not randomized to placebo treatment during chronic period, with treating the missing data as non-responders.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 200 mg -> PF-06651600 50 mg | Placebo -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg
Number analyzed (Participants) | 12 | 46 | 42 | 44 | 11 | 42 | 41 | 41
Percentage of participants | 16.7 [4.5 to 39.8] | 23.9 [15.1 to 35.0] | 28.6 [17.4 to 41.0] | 34.1 [22.3 to 46.5] | 18.2 [4.9 to 43.6] | 21.4 [12.6 to 34.2] | 26.8 [17.1 to 39.8] | 26.8 [17.1 to 39.8]

35. Secondary Outcome: Percentage of Participants Achieving Improvement in Endoscopic Appearance Based on Mayo Score at Week 32 (Chronic Period)
Description: The Mayo Score is a tool designed to measure disease activity for ulcerative colitis. The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores, which are stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscore graded 0 to 3 with the higher score indicating more severe disease activity. Improvement in endoscopic appearance was defined at Mayo endoscopic subscore of ≤1.
Time Frame: Week 32
Population: as for outcome 34
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 200 mg -> PF-06651600 50 mg | Placebo -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg
Number analyzed (Participants) | 12 | 46 | 42 | 44 | 11 | 42 | 41 | 41
Percentage of participants | 33.3 [15.4 to 60.2] | 26.1 [15.8 to 37.7] | 40.5 [27.7 to 54.3] | 34.1 [22.3 to 46.5] | 18.2 [4.9 to 43.6] | 31.0 [19.4 to 43.3] | 34.1 [23.0 to 46.9] | 36.6 [24.6 to 50.0]

36. Other Pre Specified Outcome: Change From Baseline in Total Mayo Score at Week 32 (Chronic Period)
Description: as for outcome 25
Time Frame: Week 32
Population: The participants with non-missing data in the MITT analysis set at Week 32. MITT analysis set that included all participants who were randomized to the study and received at least one dose of the randomized investigational drug, but were not randomized to placebo treatment during chronic period.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 200 mg -> PF-06651600 50 mg | Placebo -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg
Number analyzed (Participants) | 10 | 39 | 36 | 35 | 9 | 39 | 38 | 37
Units on a scale | -4.88 [-6.19 to -3.57] | -5.54 [-6.26 to -4.82] | -5.55 [-6.24 to -4.85] | -6.12 [-6.83 to -5.41] | -4.45 [-6.45 to -2.45] | -5.26 [-6.12 to -4.39] | -5.21 [-6.09 to -4.32] | -5.44 [-6.39 to -4.48]

ADVERSE EVENTS:
Time Frame: From the time the participants took at least 1 dose of study treatment up to 28 days after the last treatment administration. (approximately 36 Weeks)
Description: The analysis of AEs included all participants who received at least one dose of PF-06651600, PF-06700841, or placebo. Totals number of participants at a higher level were not necessarily the sum of those at the lower levels since a participant may report two or more different AEs within the higher level category.
Arm/Group | Placebo (Induction) | PF-06651600 20 mg (Induction) | PF-06651600 70 mg (Induction) | PF-06651600 200 mg (Induction) | PF-06700841 10 mg (Induction) | PF-06700841 30 mg (Induction) | PF-06700841 60 mg (Induction) | PF-06651600 200 mg -> PF-06651600 50 mg | PF-06651600 70 mg -> PF-06651600 50 mg | PF-06651600 20 mg -> PF-06651600 50 mg | Placebo -> PF-06651600 50 mg | PF-06700841 60 mg -> PF-06700841 30 mg | PF-06700841 30 mg -> PF-06700841 30 mg | PF-06700841 10 mg -> PF-06700841 30 mg | Placebo -> PF-06700841 30 mg | Pooling Placebo During Chronic
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/51 | 0/49 | 0/50 | 0/48 | 0/47 | 0/47 | 0/35 | 0/36 | 0/39 | 0/10 | 0/38 | 0/37 | 0/39 | 0/9 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/25 | 3/51 | 0/49 | 3/50 | 1/48 | 3/47 | 1/47 | 3/35 | 1/36 | 1/39 | 0/10 | 2/38 | 4/37 | 2/39 | 0/9 | 0/37
Other Adverse Events (participants affected / at risk) | 4/25 | 8/51 | 6/49 | 5/50 | 2/48 | 11/47 | 9/47 | 9/35 | 21/36 | 11/39 | 8/10 | 15/38 | 15/37 | 20/39 | 4/9 | 15/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Induction) (N=25) | PF-06651600 20 mg (Induction) (N=51) | PF-06651600 70 mg (Induction) (N=49) | PF-06651600 200 mg (Induction) (N=50) | PF-06700841 10 mg (Induction) (N=48) | PF-06700841 30 mg (Induction) (N=47) | PF-06700841 60 mg (Induction) (N=47) | PF-06651600 200 mg -> PF-06651600 50 mg (N=35) | PF-06651600 70 mg -> PF-06651600 50 mg (N=36) | PF-06651600 20 mg -> PF-06651600 50 mg (N=39) | Placebo -> PF-06651600 50 mg (N=10) | PF-06700841 60 mg -> PF-06700841 30 mg (N=38) | PF-06700841 30 mg -> PF-06700841 30 mg (N=37) | PF-06700841 10 mg -> PF-06700841 30 mg (N=39) | Placebo -> PF-06700841 30 mg (N=9) | Pooling Placebo During Chronic (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Listeria encephalitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Induction) (N=25) | PF-06651600 20 mg (Induction) (N=51) | PF-06651600 70 mg (Induction) (N=49) | PF-06651600 200 mg (Induction) (N=50) | PF-06700841 10 mg (Induction) (N=48) | PF-06700841 30 mg (Induction) (N=47) | PF-06700841 60 mg (Induction) (N=47) | PF-06651600 200 mg -> PF-06651600 50 mg (N=35) | PF-06651600 70 mg -> PF-06651600 50 mg (N=36) | PF-06651600 20 mg -> PF-06651600 50 mg (N=39) | Placebo -> PF-06651600 50 mg (N=10) | PF-06700841 60 mg -> PF-06700841 30 mg (N=38) | PF-06700841 30 mg -> PF-06700841 30 mg (N=37) | PF-06700841 10 mg -> PF-06700841 30 mg (N=39) | Placebo -> PF-06700841 30 mg (N=9) | Pooling Placebo During Chronic (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 4 | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 5 | 3 | 1 | 1 | 0 | 0 | 4 | 5 | 2 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1 | 3 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 4 | 0 | 1
Headache (Nervous system disorders) | 2 | 3 | 3 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 4 | 3 | 2 | 2 | 6 | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 1
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 3 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT02958865/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT02958865/SAP_001.pdf